CLINICAL TRIAL: NCT01947166
Title: Pancreatic Resection, Malnutrition, and Readmission: Assessment and Prevention
Brief Title: Pancreatic Resection, Malnutrition and Readmission
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00047214
Record Dates: First submitted 2013-08-23; First posted 2013-09-20 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Pancreatic Cancer; Malnutrition
Keywords: Whipple
MeSH Terms: conditions — Pancreatic Neoplasms; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Nestle Impact Advanced Recovery nutritional supplement — Before Surgery: Consume 1 drink box (8 ounces) three times a day for 5 days (15 servings total) on postoperative day minus 5 through postoperative day 1 in addition to normal diet. After Surgery: Consume 1 drink box (8 ounces) three times a day for 5 days on postoperative day 2 through postoperative day 6.

SUMMARY:
The Whipple procedure is associated with increased readmission rates for infection, pancreatic leak, and failure to thrive/malnutrition. The purpose of this study is to develop an evidence based perioperative nutrition plan to improve patient outcomes. The study has two specific aims including evaluation of feasibility of implementing an evidence based perioperative nutritional plan for patients undergoing Whipple and evaluation of impact of a standard perioperative nutritional plan on primary outcome of readmission rate and secondary outcomes of readmission cause, length of stay for initial hospitalization and/or readmission, post surgical complications (surgical site infections, pancreatic leak, sepsis, delayed gastric emptying), and nutritional status (PG-Subject Generated Assessment scores, BMI, albumin, pre-albumin, and method of oral intake). Categorical variables including readmission rate, readmission cause, post-surgical complications and nutritional status will be compared by chi-square test between intervention and control group. Length of stay for initial hospitalization and readmission will be compared by non parametric Wilcoxon test between two groups. Descriptive statistics will be used to describe the sample. There are no risks to the study participants.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years of age)at Duke Cancer Center
* Malignant pancreatic disease, undergoing surgical resection with pancreaticoduodenectomy (Whipple)
* Able to read and speak English.

Exclusion Criteria:

* Patients receiving preoperative enteral nutrition
* Inability to tolerate preoperative oral intake

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of implementing an evidence based perioperative nutritional plan for patients undergoing Whipple as measured by percentage of adherence to nutritional protocol | Up to week 6
  Evaluate the feasibility of implementing an evidence based perioperative nutritional plan for patients undergoing Whipple by outcomes of: 1)admission rates, 2) admission causes 3)percentage of adherence to nutritional protocol 4) length of stay 5) reported symptoms (nausea, vomiting, diarrhea), 6) postsurgical complications 7) nutritional status preoperative visit between days 2 - 5 postoperatively, on the day of discharge, and at follow up visits at weeks 1, 3 and 6.
Readmission Rate | Up to week 6
  Evaluate the impact of a standard perioperative nutritional plan on primary outcome of readmission rate.

SECONDARY OUTCOMES:
Readmission cause | Up to week 6
  Evaluate the impact of a standard perioperative nutritional plan on readmission cause.
Length of stay for initial hospitalization and/or readmission | Up to week 6
  Evaluate the impact of a standard perioperative nutritional plan on length of stay for initial hospitalization and/or readmission.
Post surgical complications | Up to week 6
  Evaluate the impact of a standard perioperative nutritional plan on post surgical complications (surgical site infections, pancreatic leak, sepsis, delayed gastric emptying) between days 2 - 5 postoperatively, on the day of discharge, and at follow up visits at weeks 1, 3 and 6.
Nutritional status | Up to week 6
  Evaluate the impact of a standard perioperative nutritional plan on nutritional status (PG-Subject Generated Assessment scores, BMI, albumin, pre-albumin, and method of oral intake) at preoperative visit, between days 2 - 5 postoperatively, on the day of discharge, and at follow up visits at weeks 1, 3 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Kara L Penne, RN, MSN, ANP, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States